CLINICAL TRIAL: NCT06013735
Title: Clinical and Microbiological Effects of Three Different Mouth Rinses Made of Sodium Fluoride, Guava Leaves Extract or Pomegranate Peel Extract on Dental Plaque in Children
Brief Title: Effects of Three Different Mouth Rinses on Dental Plaque in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 241/2019
Record Dates: First submitted 2023-07-08; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2021-09

CONDITIONS: Gingival Diseases
MeSH Terms: conditions — Gingival Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- sodium fluoride solution (Active Comparator): children will rinse with sodium fluoride solution mouth rinse (0.2%).
  Interventions: Drug: sodium fluoride solution
- guava leaves (Active Comparator): children will rinse with guava leaves aqueous extract mouth rinse (0.5%).
  Interventions: Drug: guava leaves aqueous extract
- pomegranate peel (Active Comparator): children will rinse with pomegranate peel aqueous extract mouth rinse (0.5%).
  Interventions: Drug: pomegranate peel aqueous extrac
- Control (Placebo Comparator): children will rinse with distilled water
  Interventions: Other: Distilled water

INTERVENTIONS:
Drug: sodium fluoride solution — sodium fluoride solution mouth rinse (0.2%).
  Arms: sodium fluoride solution
Drug: guava leaves aqueous extract — guava leaves aqueous extract mouth rinse (0.5%)
  Arms: guava leaves
Drug: pomegranate peel aqueous extrac — pomegranate peel aqueous extract mouth rinse (0.5%).
  Arms: pomegranate peel
Other: Distilled water — placebo distilled water
  Arms: Control

SUMMARY:
Dental plaque is a major problem in the field of oral and dental health and its prevention is more important to avoid dental caries and gingival diseases. Mouth washes are very useful in the reduction of microbial plaque and gingival inflammation. Sodium fluoride mouth wash is one of the ways that prevent dental plaque. Recently, using herbal products are efficient in decreasing dental plaque. Pomegranate peels and Guava leaves extracts are an essential medicinal plant with various pharmacological properties.

Aim of study: To evaluate and compare the efficiency of different mouth rinses (sodium fluoride mouth rinse, guava leaves aqueous extract and pomegranate aqueous extract) on dental plaque in children, clinically by measuring gingival and plaque indices scores and microbiologically by measuring of streptococcus mutans and lactobacillus.

Materials and methods: forty apparently healthy and cooperative children were selected from the Outpatient Dental Clinic of Pediatric dentistry Department, Faculty of Dentistry, Suez Canal University. Children were randomly divided into three groups as follows:

Group (I):10 children will rinse with sodium fluoride, Group (II): 10 children will rinse with guava leaves aqueous extract and Group (III):10 children will rinse with pomegranate peels aqueous extract. Group (IV):10 children will rinse with water (control group). Instructions for oral hygiene and using mouth wash will be demonstrated for every child. Clinical and microbiological examinations will be done firstly at day one before using any type of examined mouthwashes (0-base line), then clinical and microbiological follow up will be done after 7 and 15 days of using different mouthwash for each group.

ELIGIBILITY:
Inclusion Criteria:

1. Children are apparently healthy.
2. Their age's ranges from 6-12 years {mixed dentition}, First permanent molars were fully erupted.
3. Children are not taking antibiotics, steroids and inflammatory therapy for two weeks before study or during this study.
4. Children are caries free at time of the study.
5. Children with no regular use of chewing xylitol gum.
6. Children without orthodontic appliance.
7. Children are not using fluoride tooth paste or any topical fluoride application at time of study.
8. Children who have dental plaque.

Exclusion Criteria:

1. Uncooperative children.
2. Children with history of allergy to dental products or their products
3. Parents refusal.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Gingival health | baseline , after 7 days and after 15 days
  gingival index score from 0 to 3, where 0 normal gingiva and 3 severe inflammation
plaque accumulation and pocket depth | baseline , after 7 days and after 15 days
  plaque index score from 0 to 3, where 0 no plaque and 3 abundance of soft matter within gingival pocket
streptococcus mutans and lactobacilli count | baseline , after 7 days and after 15 days
  calculate the counts of streptococcus mutans and lactobacilli

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry Suez canal university, Ismailia, Egypt